CLINICAL TRIAL: NCT01233583
Title: Enumeration and Functional Evaluation of Regulatory T-cells in Psoriasis Patients Before and After Treatment With: Calcipotriol/Betamethasone, Acitretin, Narrow-Band UVB and Anti-TNF Alpha Therapy (Etanercept, Adalimumab and Infliximab)
Brief Title: Regulatory T-cells in Psoriasis Patients as Targets for Therapy
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: pRGF/009/10
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Psoriasis
Keywords: Regulatory T-cells, psoriasis, IL-10.
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination; Acitretin; Etanercept

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood Skin biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Betamethasone/Calcipotriol (Dovobet): patients in whom decision to treat with Dovobet by their dermatologist
  Interventions: Drug: Dovobet, neotigason, etanercept, adalimumab. infliximab
- Acitretin (neotigason): patients in whom decision to treat with neotigason by their dermatologist
  Interventions: Drug: Dovobet, neotigason, etanercept, adalimumab. infliximab
- narrow-band UVB: patients in whom decision to treat with narrow band UVB by their dermatologist
  Interventions: Drug: Dovobet, neotigason, etanercept, adalimumab. infliximab
- Anti TNF-alpha: patients in whom decision to treat with anti TNF-alpha(adalimumab-etanercept-infliximab) by their dermatologist
  Interventions: Drug: Dovobet, neotigason, etanercept, adalimumab. infliximab

INTERVENTIONS:
Drug: Dovobet, neotigason, etanercept, adalimumab. infliximab — Dovobet ointment 15g/day for 6 weeks Neotigason capsule 50mg per day (oral) for 6 weeks Enbrel 50mg twice weekly subcutaneous injection for 6 weeks Humira 80mg week 0, 40 mg week 1 then every other week therafter subcutaneous injection for 6 weeks Remicade 3 separate doses of 5mg/kg intavenous injection for 6 weeks

SUMMARY:
The aim of this study is to understand which therapies will suppress effector cells and promote regulatory T cells and To test whether patients with a better response to therapy and longer psoriasis-free periods develop a higher numerical ratio of regulatory to effectors T-cells and/or regulatory cells more able to suppress the effectors.

DETAILED DESCRIPTION:
This is an observational study for the effect of different treatment options of psorisis on regulatory T-cells. Patients in whom a decision to treat with one of the following therapies (Dovobet, neotigason, narrow-band UVB and anti TNF alpha therapy) and agreed to take part in the study will be selected. Allocation of different treatments to patients is not part of the study. We will enroll 40 patients with moderate to severe psoriasis in the age range from 18 to 70. patients must be treatment-free for at least 2 weeks for topical application and 4 weeks for systemic treatment of psoriasis. females of child bearing potential must be on reliable contraception. Children below 18 years, patients above 70 years, pregnant and lactating patients and immunosuppressed patients are excluded from this study. Blood and tissue samples will be taken before and after treatment. We will also invite 10 patients who are receiving ellipse excisions of naevi, and who known not to have psoriasis, to provide control samples of distal skin beyond the margins required to demonstrate complete removal and control donation of blood.

ELIGIBILITY:
Inclusion Criteria:

* • Male and female patients in the age range from 18 to 70 who are diagnosed with moderate to severe psoriasis.

  * Patients must be treatment free for at least 2 weeks for topical application and 4 weeks for systemic treatment of psoriasis.
  * Women of child bearing potential must be on reliable contraception.
  * Patients in whom a decision to treat with one of the following therapies has already been made based on normal clinical care:

    * Dovobet
    * Neotigason
    * Narrow-band UVB
    * Etanercept
    * Adalimumab
    * Infliximab
  * 10 normal controls

Exclusion Criteria:

* • Children below 18 years and patients over 70 years.

  * Pregnant and lactating patients.
  * Patients who are known to have immunosuppressive disease (e.g. HIV) or on any immunosuppressive therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and control in this study will be identified and recruited from the department of Dermatology by clinical members of the study team.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Clincal-immunological correlation of treatment outcome in psoriasis patients | 12 months
  Primary outcome measures will be the first correlations of treatment outcome in psoriasis patients assessed by PASI score and PGA, with changes in the balance between Treg and effector T cells. This will test whether changes to this balance should be a major target for future therapies. In the short term, the results will also determine whether the balance provides a useful predictive biomarker for response to treatment. It is anticipated that the results will be disseminated through publications in high impact journals and presentation at relevant scientific and clinical meetings

CONTACTS AND LOCATIONS:
Overall Officials: Anthony D Ormerod, Consultant, Principal Investigator — University of Aberdeen & NHS Grampian
Locations (1):
- Burnside House, Aberdeen, United Kingdom